CLINICAL TRIAL: NCT04528940
Title: Correlation Between Grade of Ovarian and Endometrial Carcinoma and the Expression of PD-1/PDL-1.
Brief Title: Tumor Grade Determines PD-1/PDL-1 Expression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWJ Barnabas Health at Jersey City Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1289969
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Endometrial Cancer; Ovarian Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PD-1/PDL-1 staining — Every endometrial or ovarian carcinoma will be stained for PD-1/PDL-1. The stage and grade of the tumor will be determined and correlation between tumor grade and stage and PD-1/PDL-1 staining will be made.

SUMMARY:
Endometrial carcinoma is the most common gynecologic cancer in the western world. Two types are usually described. Type I is the endometrioid and is usually estrogen dependent. Type II is usually more aggressive than type I and is estrogen independent. Type II endometrial cancer is usually characterized as high grade while type I as low intermediate and high grade. Ovarian carcinoma as opposed to endometrial carcinoma is not characterized by types but by different histological backgrounds. It is also divided into high and low grade tumors. Ovarian carcinoma is considered to be the most aggressive of all gynecological malignancies resulting in most yearly deaths. Our immune system usually responds to foreign intruders entering our body or formed inside and attacks it in order to destroy it. Cancer cells are considered to be foreign to the body hence the immune system is expected to destroy it . The immune mediated cells which are supposed to attack the cancer are called tumor infiltrating lymphocytes or "TILS". Many different cancers possess the ability to evade TILS in order to survive and grow. Many studies have demonstrated that the presence of large number of TILS improved cancer prognosis. One of these evasive methods is the PD-1/PDL-1 expression. The question whether more aggressive tumors possess better capabilities to evade an immune response via the PD-1/PDL-1 mechanism is currently unknown. All tumor types possess antigens on their cell surface which triggers an immune response to some extent. Even though, the tumor needs different methods in order to be able to avoid the immune system attack. TILS express the PD-1 receptor on their cell surface and when it binds to PDL-1 or PDL-2, the cells which express the ligand deactivate TILS hence deem the lymphocyte incapable of inducing programmed cell death. PDL-1 which is expressed on tumor cells to evade an immune response can be targeted by immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

All ages Endometrial carcinoma Ovarian carcinoma All grades All stages All races Female patients PD-1/PDL-1 staining positive -

Exclusion Criteria:

Any cancer which is not endometrial or ovarian Cancer which do not stain positive for PD-1/PDL-1

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female genital tract specific carcinomas
Study Population: The sample consists of 100 patients from all ages and races. These patients have to be diagnosed with either ovarian or endometrial carcinoma of all stages and grades. In addition, the cancerous specimen needs to stain positive for PD-1/PDL-1.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-25 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between tumor grade and prevalence of PD-1/PDL-1 histologic staining | Through study completion, an average of 12 months
  The purpose of the study is to show that the more the tumor is aggressive the higher is the prevalence of PD-1/PDL-1 staining. so every endometrial and ovarian tumors diagnosed will be stained and linear regression curves constructed to look for correlation

CONTACTS AND LOCATIONS:
Overall Officials: ariel polonsky, Principal Investigator — Jersey city medical centers
Locations (1):
- Jersey city medical center, Jersey City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided